CLINICAL TRIAL: NCT04999046
Title: A Pilot, Single Blind, Randomized Crossover Study to Evaluate the Safety and Efficacy of NaviFUS™ System Neuromodulating Treatment for Patients With Drug Resistant Epilepsy
Brief Title: NaviFUS™ System Neuromodulating Treatment for Patients With Drug Resistant Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NaviFUS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NF-2021-01
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FUS treatment (Experimental): FUS treatment will be conducted with following exposure parameters: intracranial spatial-peak temporal-average intensity (ISPTA) ceiling level: 2.8 W/cm2 (the focused ultrasound intensity in brain area considering transcranial attenuation), burst length: 3 ms, duration: three consecutive 5-minute FUS exposures with two 5-minute intermission intervals. The FUS exposure area will be the epileptogenic focus which is individually different and determined by standard clinical practice previously.
  Interventions: Device: NaviFUS System
- Sham treatment (Sham Comparator): Sham treatment is to mimic the FUS treatment procedure but without any energy. The ISPTA will be 0 W/cm2, duration: three repeating 5-minute sham exposures with two 5-minute intermission intervals.
  Interventions: Device: NaviFUS System

INTERVENTIONS:
Device: NaviFUS System — FUS treatment will be conducted with following exposure parameters: intracranial spatial-peak temporal-average intensity (ISPTA) ceiling level: 2.8 W/cm2 (the focused ultrasound intensity in brain area considering transcranial attenuation), burst length: 3 ms, duration: three consecutive 5-minute FUS exposures with two 5-minute intermission intervals.

SUMMARY:
To evaluate the safety and efficacy of using NaviFUS™ system in patients with drug resistant epilepsy

DETAILED DESCRIPTION:
This is a pilot, single blind, randomized crossover design, and single center. DRE patients with a determined epileptogenic foci will be enrolled. After completing the informed consent, patients will enter the 28-day screening period for baseline observation. Patients who had at least 3 seizures during the screening period will be eligible to participate the clinical trial. Eligible patients will be randomized into two groups to receive Sham treatment or FUS treatment on day 1. After FUS/Sham treatment, patients will be under home monitor to record the seizure by daily diary card for 1 month. After 1 month (Day 30±7), patients will be crossed over to the other treatment. Another one month observation will be necessary. In this trial, patients will totally receive 2 treatments: one FUS treatment, and one Sham treatment. Sixty (±7) days after day 1, patients will have a follow-up visit and overall evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥20 years old.
2. Patients with drug-resistant epilepsy (defined as at least 3 ASM failed) and 1-4 ASM at the time of study entry.
3. An epileptogenic foci is determined by comprehensive presurgical evaluation
4. Seizure number is countable and had been recorded at least 6 times within 2-month in medical history before screening period.
5. Seizure number had been recorded at least 3 times within 28-day screening period.
6. Willing and able to sign written informed consent and be able to comply with the study protocol during the study period.

Exclusion Criteria:

1. Patients with concurrent active psychiatric or mood disorders that in the opinion of the investigator would interfere with participation in the study.
2. Presence of pacemaker, implantable cardioverter-defibrillator (ICD), permanent medication pumps, cochlear implants, or deep brain stimulation (DBS)
3. The skull bone area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp.
4. Clips or other metallic implanted objects in the FUS exposure path, except shunts.
5. Abnormal coagulation profile:

   1. Platelet (PLT) < 100,000/μL.
   2. prothrombin time (PT) >14 sec.
   3. activated partial thromboplastin time (APTT) >36 sec.
   4. and international normalized ratio (INR) > 1.3.
6. Pregnant or breast-feeding women.
7. Coexisting medical problems of sufficient severity to limit compliance with the study.
8. Known sensitivity/allergy to Magnetic Resonance Imaging (MRI) contrast agents or any of its components.
9. Use of any recreational drugs or history of drug addiction or known history of substance or alcohol abuse.
10. Patients have received an investigational drug or an investigational device within 4 weeks prior to the study.
11. Any other condition that, in the investigator's judgment, might affect study endpoints or might increase the risk to the patients or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.
12. Any ASM treatment change during the baseline (screening period)
13. Vagus nerve stimulation (VNS) dosing changes within 2 months before baseline (screening period).
14. Radiofrequency thermocoagulation (RFTC) within 2 months before baseline (screening period).
15. Any other condition that, in the investigator's judgment, patient not applicable to participate this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Safety during study period using the NaviFUS™ System in drug resistant epilepsy patients | up to 2 months
  The number and severity of adverse events

SECONDARY OUTCOMES:
Seizure frequency | up to 2 months
  seizure diary will be utilized during long-term (two months) home monitoring and the recording will be analyzed.
Responder rate | up to 2 months
  seizure diary will be utilized during long-term (two months) home monitoring and the recording will be analyzed.
Quality of Life in Epilepsy (QOLIE-31) | up to 2 months
  A survey of health-related quality of life with epilepsy.
Number of seizure-free days | up to 2 months
  seizure diary will be utilized during long-term (two months) home monitoring and the recording will be analyzed.
Beck Anxiety Inventory (BAI) | up to 2 months
  common symptoms of anxiety
Beck Depression Inventory (BDI) | up to 2 months
  To survey patient's feeling

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No